CLINICAL TRIAL: NCT06455007
Title: Propolis as a Treatment Option for Hand Foot and Mouth Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Murat Sutcu (Other)
Responsible Party: Sponsor-Investigator, Murat Sutcu, Clinical Professor, Eskisehir Osmangazi University
Organization: Eskisehir Osmangazi University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMFD-24
Record Dates: First submitted 2024-05-31; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Children Diagnosed With HMFD; Propolis Antiviral Activity
Keywords: HMFD; children; Propolis
MeSH Terms: interventions — Propolis

STUDY DESIGN:
Intervention Model Description: control and treatment group
Masking Description: Patients in both groups were prescribed antipyretics and antihistamines when deemed appropriate by the clinician. Propolis 3x10 drops (7 days) were used in the propolis group. Both the investigators and the patients were aware of the drug being given.
  A computerized randomization program was used for group selection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propolis group (Experimental): . Propolis 3x10 drops (7 days) were used in the propolis group.
  Interventions: Drug: Propolis
- Control group (No Intervention)

INTERVENTIONS:
Drug: Propolis — Propolis 3x10 drops (7 days)
  Arms: Propolis group

SUMMARY:
Hand foot and mouth disease (HFMD) is a frequently self-limited viral infectious disease in children with no specific antiviral treatment option. There has been an increasing interest in bee products in recent years, and propolis has come to the fore with its high therapeutic and protective effect. Although the inhibitory effect of propolis against enteroviruses (EVs) has been shown in studies, there is no clinical data regarding its use in the course of HFMD.

The aim of this prospective multicenter randomized clinical study was to evaluate the effect of propolis use in children with HFMD. The patients were randomly assigned to have Anatolian propolis or no supplement - control group in addition to symptomatic therapy decided by the physician. The duration of the patients' complaints, the distribution of the lesions in the body, and the fever status were recorded on admission. Parents were asked to rate the severity of the child's restlessness, inappetence, and sleeplessness status on a scale of 0-10 on the initial, 2nd (at 48th hour), and 3rd (on 5-7 days) visits.

DETAILED DESCRIPTION:
Title of the Research Project / Thesis: "Evaluation of the effectiveness of Propolis in children with hand, foot and mouth disease"

INTRODUCTION AND PURPOSE Hand, foot and mouth disease is a highly contagious viral disease, especially in children under 10 years of age. Rarely, the disease can also be seen in older children and adults. It is a clinical picture characterized by fever, sore throat, loss of appetite, weakness, and rashes in and around the mouth, palms and soles of the feet. Rashes can be in the form of red, round lesions, or sometimes they can be seen in the form of fluid-filled vesicles. Hand, foot and mouth disease is mostly a self-limiting viral disease that does not cause severe disease. Patients recover completely within 7 to 10 days with the disappearance of all developing findings. As a very rare complication, it can cause viral or aseptic meningitis.

The patients were planned to be divided into two groups by randomization, the propolis group and the placebo group. Fever, sore throat, loss of appetite, weakness, rash and other complaints of the patients will be recorded at the time of admission and treatment will be started according to the randomization group. The patient will be given a family follow-up form and will be asked to follow up the complaints. At the 48th and 72nd hours of the follow-up, the patient was scheduled to be called for the first follow-up in terms of complaints and undesirable effects. The second and final follow-up was planned to be done on the 10th day and the patient follow-up was terminated as a family follow-up card. The number of patients targeted to be reached was determined as 100 for each group. The study period is foreseen as a total of 12 months, including 6 months for the collection of samples and data, 6 months for statistical analysis, evaluation of the results and writing them as an article. Statistical evaluation of the findings will be made with a statistical package program.

DOSES; Propolis 3x5 drops

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HMFD
* 1-10 years old

Exclusion Criteria:

* The patients whose complaints were longer than 48 hours,
* those whose parents stated that they could not comply with the follow ups,
* those who were taking another antiviral or supportive treatment,
* those who had used antibiotics in the last 1 month,
* those with a history of immunodeficiency or a family history of immunodeficiency,
* those who had a history of anaphylaxis with any support product or drug,
* patients with a chronic disease or skin lesion

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Propolis treatment | 48 hours and 7 days
  Parents were asked to rate the severity of the child's restlessness, inappetence, and sleeplessness status on a scale of 0-10. The patients' fever status, restlessness, inappetence, and sleeplessness scores were asked again to their parents and recorded. total duration of the disease and the duration of restlessness, inappetence, and sleeplessness were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University Medicine Faculty Hospital, Esenyurt, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Yes, ıt will be shared after publication.